CLINICAL TRIAL: NCT03964298
Title: Study of the Activity of PD-1 Inhibitors in Metastatic Uveal Melanoma
Acronym: imMUno
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC-2016-05
Record Dates: First submitted 2017-07-12; First posted 2019-05-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biocollection of tumoral tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study of the activity of PD-1 inhibitors in metastatic uveal melanoma

DETAILED DESCRIPTION:
The aim of the research is to study the activity of PD-1 inhibitors in patients with metastatic uveal melanoma and treated by Nivolumab and Pembrolizumab. These molecules have already received the authorities approvals. The data collected will be crucial for the understanding of the mechanism of PD-1 inhibitors and also for the futures studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic uveal melanoma
* Patients who received at least once injection of Nivolumab or Pembrolizumab in the case of the disease's treatment

Exclusion Criteria:

* Antecedent of another evolutionary tumor pathology

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic uveal melanoma.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Response rate Data collection of the efficacity of PD-1 inhibitors | December 2019
  Description of Response rate
Progression Free Survival Data collection of the efficacity of PD-1 inhibitors | December 2019
  Description of PFS (Progression Free Survival)
Global Survival Data collection of the efficacity of PD-1 inhibitors | December 2019
  Description of Global Survival
Stability Data collection of the efficacity of PD-1 inhibitors | December 2019
  Description of Stability at 6 months
Objective response Data collection of the efficacity of PD-1 inhibitors | December 2019
  Description of Objective response

SECONDARY OUTCOMES:
Exploration of PD-1 inhibitors biomarkers | December 2019
  The study of PD-1 inhibitors biomarkers could be useful to identify a group of patients whose the molecules are most activated and then for futures studies.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodrigues, MD, Study Director — Institut Curie
Locations (1):
- Rodrigues, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saint-Ghislain M, Derrien AC, Geoffrois L, Gastaud L, Lesimple T, Negrier S, Penel N, Kurtz JE, Le Corre Y, Dutriaux C, Gardrat S, Barnhill R, Matet A, Cassoux N, Houy A, Ramtohul T, Servois V, Mariani P, Piperno-Neumann S, Stern MH, Rodrigues M. MBD4 deficiency is predictive of response to immune checkpoint inhibitors in metastatic uveal melanoma patients. Eur J Cancer. 2022 Sep;173:105-112. doi: 10.1016/j.ejca.2022.06.033. Epub 2022 Jul 19. PMID 35863105